CLINICAL TRIAL: NCT03086005
Title: A Multicenter, Prospective, Randomized Study to Assess the Effect of Metformin Supplementation on IVF Outcome and Intrafollicular Environment in Patients With Polycystic Ovarian Syndrome Undergoing In Vitro Fertilization/Embryo Transfer
Brief Title: Study to Assess the Effect of Metformin Supplementation on IVF Outcome in Patients With Polycystic Ovarian Syndrome.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chung-Hoon Kim (Other)
Responsible Party: Sponsor-Investigator, Chung-Hoon Kim, Asan Medical Center, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-Metformin for PCOS
Record Dates: First submitted 2017-02-15; First posted 2017-03-22 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Metformin
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): Metformin 500mg tablet by mouth, every 12 hours, from the first day of oral contraceptive pills taken to the day of oocyte retrieval
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo(identical in appearance to metformin), every 12 hours, from the first day of oral contraceptive pills taken to the day of oocyte retrieval
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin
  Other Names: Glucophage Tab 500mg, National Drug Code(NDC) 0087-6060-05

SUMMARY:
This study was performed to investigate the effects of metformin on controlled ovarian stimulation (COS), in vitro fertilization (IVF) outcomes, pregnancy outcomes, and comparison of serum and follicular fluid cytokines and hormones in patients with polycystic ovary syndrome (PCOS) undergoing IVF using gonadotropin-releasing hormone(GnRH) antagonist protocol.

DETAILED DESCRIPTION:
Polycystic ovary syndrome is the common cause of the female infertility that features insulin resistance and hyperinsulinemia participate in the reproductive as well as metabolic disturbances.

In many studies, metformin treatment reduces androgen levels and attenuates hyperinsulinemia in women with PCOS. This favorable effect on insulin and androgens levels, justifies the use of metformin in reproductive disturbances in PCOS women. Metformin treatment was shown to diminish ovarian androgen secretion, while lowering insulin levels in women with PCOS.

In women with PCOS, metformin treatment may increase ovulation, improve menstrual cyclicity, and reduce seum androgen levels. Metformin has direct effects on the ovary and also reduces the level of insulin that act upon the ovary. It has been indicated that metformin has direct, insulin-independent actions on theca cell steroidogenesis, because in human ovarian theca-like tumor cells, metformin suppressed androstenedione production. Metformin also exert a direct effect on granulosa cells and subsequent reduction of steroid production.

Metformin was shown to improve endothelium dependent vasodilation in insulin resistant patients and potentially protect against atherogenesis and cardiovascular disease.

Considering gonadotropin ovulation induction or IVF in women with PCOS, metformin coadministration improves the pregnancy outcome and reduces the risk of ovarian hyperstimulation syndrome. Metformin therapy throughout pregnancy can reduce the risk of early miscarriage or the incidence of gestational diabetes.

All patients were pretreated for 3 weeks with monophasic oral contraceptive (OC)(Yasmin; Bayer Schering Pharma, Berlin, Germany) before COS. Five days after OC discontinuation, COS for IVF/ICSI was commenced. GnRH antagonist protocol was used for COS in all subjects. Patients were randomly allocated into the metformin or control groups, using sealed envelopes.

ELIGIBILITY:
Inclusion Criteria:

* PCOS diagnostic criteria

  * 2003 American Society for Reproductive Medicine(ARSM)/European Society of Human Reproduction and Embryology(ESHRE) consensus meeting guideline
  * include two out of three

    1. Oligo - or anovulation
    2. Clinical or/and biochemical hyperandrogenism
    3. Polycystic ovaries on ultrasound, exclusion of other etiologies( ≥ 12 follicles(2-9 mm diameter) in each ovary or ovarian volume(0.5 x length x width x thickness) ≥ 10cm3)
* Anatomical normal uterus
* Normal level of thyroid hormone

Exclusion Criteria:

* Severe endometriosis(stageIII, IV)
* Endometrial thickness less than 7mm in late follicular phase
* Severe male infertility factor, non-obstructive azoospermia
* History of ectopic pregnancy or abortion over the last 3 months
* Unexplained abnormal uterine bleeding
* Congenital adrenal hyperplasia
* Androgen secreting tumor
* Cushing syndrome
* Concurrent administration of metformin, ovulation induction drugs, oral contraceptives within previous 3 months
* Chronic disease(liver, kidney, severe heart failure, DM)
* Any pathology of genital tract
* History of alcohol abuse
* Refuse of study participate consent

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10-12 (Actual); Primary Completion 2015-05-04 (Actual); Study Completion 2015-07-23 (Actual)

PRIMARY OUTCOMES:
Number of mature(MII) oocyte | Day1(from the day of oocyte retrieval to fertilization confirmation)
  using polarized light microscopy

SECONDARY OUTCOMES:
Clinical pregnancy rate in % | Pregnancy test was carried out at 11 days after embryo transfer and was classified as positive when the serum beta-human chorionic gonadotropin(hCG) level was over 5 IU/L. Than follow up to 12 weeks of gestation.
  Clinical pregnancy was defined as a viable pregnancy beyond 12 weeks gestation by ultrasonographic visualization.
Miscarriage rate in % | Pregnancy test was carried out at 11 days after embryo transfer and was classified as positive when the serum beta-human chorionic gonadotropin(hCG) level was over 5 IU/L. Than follow up to 20 weeks of gestation.
  Miscarriage was defined as a early loss of a pregnancy before 20 weeks of pregnancy.
Total dose of follicle-stimulating hormone(FSH) used(IU) | average of 10 days, From the day of stimulation start with FSH to the day of oocyte retrieval
  compare the ovarian response to controlled ovarian stimulation between two groups
Total duration of FSH used(day) | average of 10 days, From the day of stimulation start with FSH to the day of oocyte retrieval
  compare the ovarian response to controlled ovarian stimulation between two groups
Number of oocytes retrieved | Day1(the day of oocyte retrieval)
  using polarized light microscopy
Number of frozen 2 pronucleus(2PN) embryos | Day1((from the day of oocyte retrieval to fertilization confirmation)
  using polarized light microscopy
Follicular fluid Tumor necrosis factor(TNF)-α level in pg/ml and follicular fluid Adiponectin level in pg/ml and follicular fluid Interleukin-6 level in pg/ml and follicular fluid Anti-mullerian hormone(AMH) level in pg/ml | Day 1
  At the day of oocyte retrieval, follicular fluids were collected from the follicles with a diameter over than 15mm. The fluids were frozen within 4 hours for the future analysis. All the samples were stored at -20℃ and were analysed in the biochemistry department of the study centre.
Serum TNF-α level in pg/ml and serum Adiponectin level in pg/ml and serum Interleukin-6 level in pg/ml and serum AMH level in pg/ml and serum Testosterone level in pg/ml and serum Estradiol level in pg/ml | Day 1
  Serum samples were obtained on the day of Metformin commencement and ovum pick up. Levels are measured by means of solid-phase enzyme-linked immunosorbent assay.

CONTACTS AND LOCATIONS:
Overall Officials: CHUNG-HUN KIM, Professor, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thessaloniki ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Consensus on infertility treatment related to polycystic ovary syndrome. Hum Reprod. 2008 Mar;23(3):462-77. doi: 10.1093/humrep/dem426. PMID 18308833
- [Background] Diamanti-Kandarakis E, Economou F, Palimeri S, Christakou C. Metformin in polycystic ovary syndrome. Ann N Y Acad Sci. 2010 Sep;1205:192-8. doi: 10.1111/j.1749-6632.2010.05679.x. PMID 20840272
- [Background] Doldi N, Persico P, Di Sebastiano F, Marsiglio E, Ferrari A. Gonadotropin-releasing hormone antagonist and metformin for treatment of polycystic ovary syndrome patients undergoing in vitro fertilization-embryo transfer. Gynecol Endocrinol. 2006 May;22(5):235-8. doi: 10.1080/14767050600761893. PMID 16785142
- [Background] Farrell K, Antoni MH. Insulin resistance, obesity, inflammation, and depression in polycystic ovary syndrome: biobehavioral mechanisms and interventions. Fertil Steril. 2010 Oct;94(5):1565-74. doi: 10.1016/j.fertnstert.2010.03.081. Epub 2010 May 14. PMID 20471009
- [Background] Katsiki N, Hatzitolios AI. Insulin-sensitizing agents in the treatment of polycystic ovary syndrome: an update. Curr Opin Obstet Gynecol. 2010 Dec;22(6):466-76. doi: 10.1097/GCO.0b013e32833e1264. PMID 20724929
- [Background] Toulis KA, Goulis DG, Farmakiotis D, Georgopoulos NA, Katsikis I, Tarlatzis BC, Papadimas I, Panidis D. Adiponectin levels in women with polycystic ovary syndrome: a systematic review and a meta-analysis. Hum Reprod Update. 2009 May-Jun;15(3):297-307. doi: 10.1093/humupd/dmp006. Epub 2009 Mar 4. PMID 19261627
- [Background] Ardawi MS, Rouzi AA. Plasma adiponectin and insulin resistance in women with polycystic ovary syndrome. Fertil Steril. 2005 Jun;83(6):1708-16. doi: 10.1016/j.fertnstert.2004.11.077. PMID 15950640
- [Derived] Tso LO, Costello MF, Albuquerque LET, Andriolo RB, Macedo CR. Metformin treatment before and during IVF or ICSI in women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2020 Dec 21;12(12):CD006105. doi: 10.1002/14651858.CD006105.pub4. PMID 33347618